CLINICAL TRIAL: NCT06825468
Title: Role Of Hysterectomy In The Treatment Of Borderline Ovarian Tumors
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HYSTEROBOT
Record Dates: First submitted 2024-12-30; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Hysterectomy
Keywords: Borderline ovarian tumours; gynaecology; perimenopause; postmenopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Borderline ovarian tumors (BOT), are rare epithelial ovarian tumors characterized by the presence of frankly malignant cytologic features in the absence of stromal invasion.

Surgical treatment of perimenopausal and postmenopausal BOT requires bilateral adnexectomy. Although some studies have reported an increased recurrence rate in the group of patients treated with uterine preservation, these data are severely limited by the small sample of patients and the presence of confounding factors in the analysis of oncologic outcomes.

Determining the impact of hysterectomy on the survival outcomes of perimenopausal and postmenopausal patients diagnosed with early FIGO stage BOT is necessary to avoid overtreatment, hysterectomy being associated with a low but not negligible rate of morbidity and mortality.

DETAILED DESCRIPTION:
Borderline ovarian tumors (BOTs), are rare epithelial ovarian tumors characterized by the presence of frankly malignant cytologic features in the absence of stromal invasion. Serous BOTs, which account for 67% of all BOTs, are limited to one ovary in 75% of cases and are frequently accompanied by predominantly noninvasive peritoneal implants. In 30% of cases, BOTs are mucinous, unilateral, and characterized by a low rate of extra-ovarian spread and invasive implants. Patients with BOT are diagnosed at FIGO stage I in 78.9% of cases, are usually young, and have a favorable prognosis with 5-year survival affecting more than 80% of patients.

Surgical treatment of perimenopausal and postmenopausal BOT requires bilateral annissiectomy. Otherwise, the role of hysterectomy in perimenopausal and postmenopausal women with early-stage BOT remains unclear. Although some studies have reported an increased recurrence rate in the group of patients treated with uterine preservation, these data are severely limited by the small sample of patients and the presence of confounding factors in the analysis of oncologic outcomes.

Determining the impact of hysterectomy on the survival outcomes of perimenopausal and postmenopausal patients diagnosed with early FIGO stage BOT is necessary to avoid overtreatment, hysterectomy being associated with a low but not negligible rate of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Women in menopause clinically defined as absence of menstrual cycle for 12 months
* Primary diagnosis of BOT confirmed by pathological examination
* Surgical treatment of BOT by BSO with (group 1) and without (group 2) hysterectomy
* Informed consent acquisition

Exclusion Criteria:

* Occurrence of BOT at index intervention
* Stage IV
* Metastatic disease
* Patients with previous hysterectomy
* Cancer synchronous of the endometrium
* Patients who have not had follow-up before 5 years (excluding those who have not reached the 5 year follow-up for the following events: death from any cause, death from BOT, recurrence of BOT)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with BOT diagnosis will be included in the study for analysis:
  * BSO and hysterectomy (group 1)
  * BSO without hysterectomy (group 2)
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Impact of uterine preservation on the rate of BOT recurrence | After surgery during follow up (up to 20 years)
  Impact of uterine preservation on the rate of borderline ovarian tumors (BOT) recurrence and thus its usefulness or otherwise in clinical care practice; therefore, the overall recurrence rate (which includes BOT, invasive BOT implants, and carcinoma) in patients treated with (group 1) and without (group 2) hysterectomy will be determined

SECONDARY OUTCOMES:
The rate of recurrence of BOT and of invasive implants | After surgery during follow up (up to 20 years)
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy the rate of recurrence of BOT and of invasive implants
The rate of carcinoma recurrence | After surgery during follow up (up to 20 years)
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy the rate of carcinoma recurrence
the overall survival (OS) defined as the time from surgery to the patient's death from any cause | After surgery during follow up (up to 20 years)
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy the overall survival (OS) defined as the time from surgery to the patient's death from any cause
disease-free survival (DFS) defined as time from surgery to recurrence | After surgery during follow up
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy disease-free survival (DFS) defined as time from surgery to recurrence
disease-specific survival (DSS) defined as the time from first surgery for BOT to death from disease | After surgery during follow up (up to 20 years)
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy disease-specific survival (DSS) defined as the time from first surgery for BOT to death from disease
the rate of postoperative complications | After surgery during follow up (up to 20 years)
  Improved care practice by determining in patients with BOT undergoing (group 1) or not undergoing (group 2) hysterectomy the rate of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma
  - Ospedale universitario, Azienda Sanitaria Universitaria Friuli Centrale, Udine